CLINICAL TRIAL: NCT00454519
Title: Cytoreductive Surgery Plus Intraoperative Peritoneal Hyperthermic Chemotherapy for the Treatment of Peritoneal Carcinomatosis From Gastrointestinal Cancer: an Open Label, Randomized, Prospective, Phase 2 Clinical Trial
Brief Title: Surgery Plus Intraoperative Peritoneal Hyperthermic Chemotherapy (IPHC) to Treat Peritoneal Carcinomatosis
Acronym: IPHC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Collaborators: NPO Organization to Support Peritoneal Dissemination Treatment (Unknown); Kishiwada Tokushukai Hospital (Other); Kusatsu General Hopital (Unknown); Ikeda Hospital (Unknown)
Responsible Party: Prof. Yan Li, M.D., Ph.D, Cancer Center of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUCC-0701
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Stomach Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Mesothelioma
Keywords: peritoneal carcinomatosis; cisplatin; mitomycin; gastric cancer; colorectal cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Mesothelioma; Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures; Cisplatin; Mitomycin; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): cytoreductive surgery, IPHC, cisplatin 20 mg/m2/L, Mitomycin C 4 mg/m2/L, postoperative chemotherapy.
  Interventions: Procedure: intraoperative peritoneal hyperthermic chemotherapy with cisplatin and mitomycin
- B (Active Comparator): cytoreductive surgery alone, postoperative chemotherapy.
  Interventions: Procedure: cytoreductive surgery

INTERVENTIONS:
Procedure: cytoreductive surgery — the whole abdominal-pelvic cavity is explored and maximal cytoreductive surgery is performed to remove visible tumor burden as much as possible.
  Arms: B
Procedure: intraoperative peritoneal hyperthermic chemotherapy with cisplatin and mitomycin — Immediately after the cytoreductive surgery, cisplatin and mitomycin C dissolved in 12,000 ml of normal saline heated to 42 degrees celsius is infused into the abdominal cavity for a sustained hyperthermic intraperitoneal chemotherapy for 60 to 90 minutes.
  Other Names: HIPEC
  Arms: A

SUMMARY:
OBJECTIVES:

* Determine response and survival of patients with peritoneal carcinomatosis treated with cytoreductive surgery plus intraoperative peritoneal hyperthermic chemotherapy with cisplatin and mitomycin
* Assess the quality of life of patients treated with this regimen.

OUTLINE: Patients are randomized into IPHC group and control group. In the former group, the patients undergo cytoreductive surgery plus intraoperative hyperthermic peritoneal perfusion with cisplatin and mitomycin over 60 minutes. Patients in the control group just underwent routine cytoreductive surgery.

All patients in both groups receive the standard conventional chemotherapy after surgery.

Quality of life is assessed at study initiation, at 1, 3, 6 months. Patients are followed at 4 weeks, every 3 months for 1 year, and then every 6 months for up to 3 years.

DETAILED DESCRIPTION:
DISEASE CHARACTERISTICS:

* Histologically confirmed peritoneal carcinomatosis with the following histologies:
* Primary peritoneal mesothelioma
* Adenocarcinoma of gastrointestinal tract origin
* Confined to peritoneal cavity
* Tumor mass could be debulked to less than 2.5 cm in diameter per tumor deposit
* Must not have failed prior intraperitoneal platinum therapy
* Treatment failure is defined as radiographic evidence of disease progression on 2 consecutive CT scans within 3 months after therapy

PATIENT CHARACTERISTICS:

Age:

- 20 to 70 years old

Performance status:

- KPS>50

Life expectancy:

- More than 8 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 80,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN
* Liver enzymes no greater than 2 times ULN

Renal:

- Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No significant irreversible cardiac ischemia
* No significant changes in ECG recording

Pulmonary:

* FEV_1 at least 1.2 liters
* Maximum voluntary ventilation at least 50% expected

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No concurrent medical problems that would preclude surgery

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer or colorectal cancer with peritoneal carcinomatosis
* Gastric cancer or colorectal cancer with malignant ascites
* Karnofsky Performance Scale(KPS)>50

Exclusion Criteria:

* Age less than 20 years old, or beyond 70 years old
* Any lung metastasis, liver metastasis, or prominent retroperitoneal lymph node metastasis
* Bilirubin greater than 3 times upper limit of normal (ULN)
* AST and ALT greater than 5 times ULN
* Liver enzymes greater than 3 times ULN

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
overall survival time | from operation to death due to cancer recurrence

SECONDARY OUTCOMES:
perioperative morbidity and mortality | Within 30 days postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, M.D., Ph.D, Principal Investigator — Cancer Center of Wuhan University; Yonemura Yutaka, MD, PhD, Principal Investigator — NPO Organization to Support Peritoneal Dissemination Treatment
Locations (1):
- Cancer Center of Wuhan University & Department of Oncology, Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Background] Yang XJ, Li Y, al-shammaa Hassan AH, Yang GL, Liu SY, Lu YL, Zhang JW, Yonemura Y. Cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy improves survival in selected patients with peritoneal carcinomatosis from abdominal and pelvic malignancies: results of 21 cases. Ann Surg Oncol. 2009 Feb;16(2):345-51. doi: 10.1245/s10434-008-0226-2. Epub 2008 Nov 19. PMID 19018599
- [Derived] Zou D, Cai Y, Jin M, Zhang M, Liu Y, Chen S, Yang S, Zhang H, Zhu X, Huang C, Zhu Y, Miao X, Wei Y, Yang X, Tian J. A genetic variant in the immune-related gene ERAP1 affects colorectal cancer prognosis. Chin Med J (Engl). 2024 Feb 20;137(4):431-440. doi: 10.1097/CM9.0000000000002845. Epub 2023 Sep 8. PMID 37690994
- [Derived] Wu HT, Yang XJ, Huang CQ, Sun JH, Ji ZH, Peng KW, Zhang Q, Li Y. Cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy with lobaplatin and docetaxel improves survival for patients with peritoneal carcinomatosis from abdominal and pelvic malignancies. World J Surg Oncol. 2016 Sep 15;14(1):246. doi: 10.1186/s12957-016-1004-4. PMID 27633880